CLINICAL TRIAL: NCT01954095
Title: Determining the Pharmacodynamic Impact of Vaginal and IM Progestins on the Cervix
Brief Title: The Impact of Vaginal and IM Progestins on the Cervix
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Indiana University (Other); University of Texas (Other); University of Washington (Other); RTI International (Other)
Responsible Party: Sponsor
Other Study IDs: OPRU Progestin
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Preterm Birth; Short Cervical Length
Keywords: 17-OHPC, Prometrium, Cerclage, Pre-term birth, Short cervix
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for DNA extraction, hormone, and metabolomic analyses
  Cervicovaginal fluid for proteome, cytokines, and matrix metalloproteins (MMPs)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1: No prior preterm birth & normal cervix length: Pregnant women at 16 0/7 - 23 6/7 weeks gestation who have had one or more term births (no prior preterm births) and have a normal cervical length (> 25 mm). These women will serve as gestational age controls for all groups.
- Group 2: No prior preterm birth & short cervix length: Pregnant women at 16 0/7 - 23 6/7 weeks gestation who have no prior preterm births and have a short cervical length (20mm or less). These women may receive treatment (e.g. vaginal progesterone, cerclage, pessary, NSAIDs, or a combination thereof) or no treatment.
- Group 3: Prior preterm birth, normal cervix length, 17-OHPC: Pregnant women at 16 0/7 - 23 6/7 weeks gestation who have had prior preterm birth, have a normal cervical length and will receive 17-OHPC treatment.
- Group 4: Prior preterm birth, normal cervix length, no treat: Pregnant women at 16 0/7 - 23 6/7 weeks gestation who have had prior preterm birth, have a normal cervical length, and will not receive any treatment. These women will serve as controls for Group 3.

SUMMARY:
The purpose of this study is to analyze how the body handles and responds to progesterone treatment in parous and nulliparous women at risk of pre-term birth.

DETAILED DESCRIPTION:
17-hydroxyprogesterone caproate (17-OHPC) has recently been shown to reduce the rate of recurrent preterm birth while intravaginal progesterone has been shown to reduce the rate of preterm birth in women with short cervix. While these interventions have reduced the rate of preterm birth, the mechanisms of action of these medications are unknown. The objective of this study is to collect and analyze blood and cervicovaginal fluids from pregnant women receiving these medications or other interventions such as cerclage, pessary, NSAIDs, and combinations thereof. The goal of the analyses is to assess the impact of these interventions on the cervical proteome, cervical cytokines and cervical structure and to identify potential biomarkers of response and non-response thus providing insights into the mechanisms of action of these drugs.

ELIGIBILITY:
Inclusion Criteria

All Groups

* Singleton gestation (16 0/7 - 23 6/7 weeks gestation)
* Willing to provide informed consent
* Age 18 - 50 years inclusive

Additionally,

Group 1: One or more prior term births (>37 0/7 weeks); No prior spontaneous birth at 16 0/7 - 36 6/7 weeks; and normal cervical length (>25 mm)

Group 2: Cervical length of 20 mm or less at 16 0/7 - 23 6/7 weeks

Groups 3 and 4: History of prior spontaneous birth at 16 0/7 - 34 0/7 weeks and normal cervical length (> 25mm) at enrollment.

Exclusion Criteria

All Groups

* Active labor
* Active bleeding
* On progestin therapy, chronic steroid, or current NSAID therapy
* Actively receiving study treatment in another clinical trial (observational trials allowed)
* Major fetal malformation lethal anomalies, or anomalies that may lead to early delivery or increased risk of neonatal death e.g., gastroschisis, spina bifida, or serious karyotypic abnormalities
* Amniotic membranes prolapsed beyond the external os (ostium of uterus) or protruding into the vagina
* Pregnancy without a viable fetus
* Prenatal care or delivery planned elsewhere (unless the study visits can be made as scheduled and complete outcome information can be obtained)

Additionally:

Group 1: Cervical dilation greater than or equal to 3cm

Group 2: Prior preterm birth (16 0/7 - 34 0/7); active deep vein thrombosis, pulmonary embolism, or history of these conditions; known liver dysfunction or disease (active hepatitis, HIV)

Group 3: inability or unwillingness to use a 17-OHPC compounded product similar in composition to the FDA-approved product; allergy to 17-OHPC or its components

Groups 1, 3, and 4: cerclage in place or anticipated; congenital mullerian abnormality of the uterus; positive for bacterial vaginosis, chlamydia, gonorrhea, or trichomonas

Groups 3 and 4: current or history of thrombosis or thromboembolic disorders; known or suspected breast cancer, other hormone-sensitive cancer, or history of these conditions; undiagnosed abnormal vaginal bleeding unrelated to pregnancy; cholestatic jaundice of pregnancy, liver tumors, benign or malignant, or active liver disease; uncontrolled hypertension

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study consists of 4 groups of women who are between 16 0/7 - 23 6/7 weeks gestation. The allocation of a subject to a group is based on two objective assessments (history of preterm birth and cervical length) and the joint clinical decision of the woman and her physician regarding treatment options.
  Study participants who have no prior preterm births and a normal cervical length will be assigned to Group 1. If the participant has no prior preterm births and a short cervical length, she will be assigned to Group 2 regardless of treatment or no treatment. Group assignment for women with a prior preterm birth and normal cervical length is based on 17-OHPC use. Participants who elect to use 17-OHPC will be assigned to Group 3 and those who choose not to receive any treatment will be assigned to Group 4.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Biomarkers | 2 Weeks
  Proteins in the cervicovaginal fluid with expression changes two-fold or greater between day 0 and week 2 of either vaginal or IM progestin therapy.

SECONDARY OUTCOMES:
Cervical sonographic changes | 8 Weeks
  Changes in cervical sonographic gray scale density/length from weeks 0-2, 0-4, and 0-8 after the start of progestin therapy.
Protein Expression | 8 Weeks
  Proteins in the cervicovaginal fluid whose expression changes significantly from weeks 0-4 and 0-8 after the start of progestin therapy.
Cervical cytokines | 8 Weeks
  Changes in cervical cytokine inflammatory ratio weeks 0-2, 0-4, and 0-8 after the start of progestin therapy.
Individual cytokines | 8 Weeks
  Changes in individual cytokines (IL-1α, IL-1β, IL-1RA, IL-4, IL-6, IL-8, IL-10, IL-13, and TNF-α) from weeks 0-2, 0-4, and 0-8 after the start of progestin therapy.
Cervical MMPs | 8 Weeks
  Changes in cervical MMPs 1, 2, 8 and 9 from weeks 0-2, 0-4, and 0-8 after the start of progestin therapy.
Single nucleotide polymorphisms | 8 Weeks
  Test for association between single nucleotide polymorphisms (SNPs) in progestin and estrogen-related candidate genes and changes in the CVF proteome and cervical density and length.
Biomarkers | 8 Weeks
  Proteins in the cervicovaginal fluid with expression changes two-fold or greater between weeks 0-4 and 0-8 of either vaginal or IM progestin therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Hebert, PharmD, FCCP, Principal Investigator — University of Washington; Steve Caritis, MD, Principal Investigator — University of Pittsburgh; Gary Hankins, MD, Principal Investigator — University of Texas; David Flockhart, MD, PhD, Principal Investigator — Indiana University School of Medicine
Locations (4):
- United States (4):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - University of Washington, Seattle, Washington